CLINICAL TRIAL: NCT02508662
Title: Registry Study for Personalized Cancer Therapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0300; NCI-2015-01453 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-07-22; First posted 2015-07-27 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Advanced Cancers; Solid Tumors
Keywords: Advanced Cancers; Solid Tumors; Genomic Mutations; FDA Approved Off-Label Chemotherapy; Refractory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (about 4 teaspoons) drawn to check for any genetic mutations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Advanced Cancer (Refractory) with Genomic Mutation: Participants with advanced cancer who have exhausted standard treatment option and have no potential clinical trial available, and who have potentially actionable alterations on genomic profiling.
  Interventions: Other: Review of Screening Tests and Molecular Test Results

INTERVENTIONS:
Other: Review of Screening Tests and Molecular Test Results — Review of screening tests and molecular test results in participant's medical records. Study staff and study doctor work together to find an off-label use for an FDA approved therapy that is best for participant.

SUMMARY:
Objectives:

Primary Objectives:

To evaluate the anti-cancer activity of commercially available, targeted anti-cancer therapies used off-label for treatment in patients with advanced solid cancer with known genomic aberrations.

Secondary Objectives:

To determine outcomes of patients who were treated with matched targeted anti-cancer therapies based on known genomic aberrations.

To obtain treatment related adverse events in patients with advanced solid tumor who were treated with off -label targeted therapies.

To determine co-genomic aberrations that may contribute to treatment response or resistance mechanisms.

To determine feasibility of detecting the genomic alterations in plasma, and the genomic evolution of circulating biomarkers.

DETAILED DESCRIPTION:
Study Treatment Assignment:

If you are found to be eligible to take part in this study, the study doctor will review the test results in your medical records that were previously performed as part of your routine care. The results of the testing may be helpful in managing your treatment and may also help the doctor to find effective off-label use of FDA approved therapies for the type of cancer you have.

After reviewing the screening tests and the molecular test results in your medical records, the study staff and your study doctor will work together to find an off-label use for an FDA approved therapy that is best for you. You may receive a single therapy or a combination of therapies. You and the study doctor will discuss this.

The study doctor or study staff will tell you which drug(s) you will be taking, the dose of the study drug(s), and how often you should take them. You will sign a separate consent form that explains in more detail how the study drug(s) are administered and the potential benefits and side effects of taking the study drug(s).

Study Visits:

While you are receiving treatment and during follow-up, you will have your routine, standard of care clinic visits and routine tests so that the doctor may check the status of the disease to learn if the therapy chosen to treat the disease is having any effect. Information from these routine visits will be collected and stored by the study staff. The timing of these visits will depend on the type of therapy you receive.

During every cycle of therapy (about every 3-4 weeks):

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If your doctor thinks it is needed, urine will be collected for routine tests.
* If your doctor thinks it is needed, you will have an EKG to check the health of your heart.

After even numbered cycles (2, 4, 6, and so on), or more often if the doctor thinks is it needed, you will have the same imaging scan(s) which were done during Screening to check the status of the disease.

This is an investigational study.

Up to 100 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced or metastatic cancer that is refractory to standard therapy or that has relapsed after standard therapy or has no standard therapy that increases survival by at least three months.
2. Patients with a potentially actionable genomic alteration.
3. All prior treatment-related toxicities must be resolved to CTCAE (Version 4.0) < or = Grade 2 (except alopecia) at the time of screening.
4. Patients willing to sign informed consent.
5. Patients under the age of 18 years old are allowed as long as the safety profile of the drug is established in the pediatric population.

Exclusion Criteria:

1. Any serious and/or unstable pre-existing medical disorder, psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures, in the opinion of the Investigator.
2. Have a known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to planned treatment drug.
3. Rapidly progressing leptomeningeal or brain metastases or spinal cord compression.
4. Clinical trial (including targeted and/or non-targeted) other than registry study is available; patient is willing and eligible to enroll in such trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with advanced solid cancer with known genomic aberrations at MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-07-21 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Tumor Response | 8 weeks
  Evaluation of tumor: the same imaging technique used during the initial evaluation or more sophisticated studies performed once after 2 cycles.
  Patients with measurable disease assessed by standard RECIST (Version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org